CLINICAL TRIAL: NCT04096066
Title: Carfilzomib - Lenalidmide - Dexamethasone (KRd) Versus Lenalidomi - Dexamethasone (Rd) in Newly Diagnosed Myeloma Patients Not Eligible for Autologous Stem Cell Transplantation: a Randomized Phas III Trial
Brief Title: A Trial That Compare Two Treatments in Newly Diagnosed Myeloma Patients Not Eligible for Transplant
Acronym: KRdvsRd
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN20
Record Dates: First submitted 2019-07-02; First posted 2019-09-19 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; New Diagnosis Tumor
Keywords: Multiple Myeloma; AUTOLOGOUS STEM CELL TRANSPLANTATION INELIGIBLE; Proteasome inhibitor; Immunomodulating agents
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- KRd (Experimental Arm) (Experimental): Carfilzomib (K):
  * 20 mg/m2 IV on day 1 of cycle 1;
  * 56 mg/m2 IV on days 8 and 15 in cycle 1;
  * 56 mg/m2 IV on days 1, 8 and 15 in cycles 2-12;
  * 56 mg/m2 on days 1 and 15 from cycle 13 and onwards.
  Lenalidomide (R):
  - 25 mg orally on days 1-21 of each cycle.
  Dexamethasone (d):
  - 40 mg orally on days 1, 8, 15 and 22 of each cycle. Each cycle is a 28-day cycle.
  Until PD or intolerance. Only patients that achieve at least a VGPR within the first year of treatment and in sustained MRD negativity (MRD negative at least at 10-5 after 1 and 2 years of therapy) will stop carfilzomib after 2 years of treatment, and will continue with lenalidomide and dexamethasone administration.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- Rd (Control Arm) (Active Comparator): Lenalidomide (R):
  -25 mg orally on days 1-21 of each cycle.
  Dexamethasone (d):
  -40 mg orally on days 1, 8, 15 and 22 of each cycle. Each cycle is a 28-day cycles.
  Until PD or intolerance.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — * 20 mg/m2 IV on day 1 of cycle 1 enhanced to 56 mg/m2 on days 8, and 15 of cycle 1;
  * 56 mg/m2 IV on days 1, 8 and 15 in cycles 2-12;
  * 56 mg/m2 IV on days 1 and 15 from cycle 13 and onwards.
  Other Names: Kyprolis
  Arms: KRd (Experimental Arm)
Drug: Lenalidomide — - 25 mg orally on days 1-21 of each cycle.
  Other Names: Revlimid
Drug: Dexamethasone — - 40 mg orally on days 1, 8, 15 and 22 of each cycle. Each cycle is to be repeated every 28 days. Patients that achieve at least a VGPR within the first year of study treatment and in sustained MRD negativity (MRD negative at least at 10-5 after 1 and 2 years of therapy) will stop carfilzomib administration after 2 years and will continue with lenalidomide and dexamethasone treatment until disease progression or intolerance to the therapy. Other patients will continue carfilzomib administration until disease progression or intolerance.
  For patients >75 years of age, the dose of dexamethasone is 20 mg/day on Days 1, 8, 15 and 22 of each treatment cycle.

SUMMARY:
The combination of lenalidomide plus low-dose dexamethasone (Rd) is considered the new standard for elderly newly diagnosed multiple myeloma (NDMM) patients. The combination carfilzomib plus lenalidomide-dexamethasone (KRd) in relapsed-refractory MM patients improved the progression-free survival (PFS) of approximately 1 year compared to standard Rd treatment. In a small phase 2 trial (23 pts) the KRd combination in elderly NDMM pts showed a complete response (CR) rate of 79% and a PFS at 3 years of 80%. Cardiovascular adverse events are the most limiting toxicities, especially in elderly patients.

DETAILED DESCRIPTION:
This protocol is a randomized, multicenter study designed to determine the MRD negativity and the PFS of KRd treatment regimen.

Patients will be randomized in a 1:1 ratio to receive carfilzomib-lenalidomide-dexamethasone (KRd - Arm A) or lenalidomide-dexamethasone (Rd - Arm B).

Patients will be stratified basing on international staging system (ISS) and fitness status using a web-based procedure completely concealed to study participants.

All consecutive patients ≥ 65 years with newly diagnosed MM will be enrolled in a large randomized study during a period of 24 months.

Patients will be treated until disease progression or intolerance to the therapy. The only exception is for patients enrolled in KRd arm who achieve at least a VGPR during the first year of treatment and in sustained MRD negativity (MRD negative at least at 10-5 after one and two years of therapy): these patients will stop carfilzomib administration after 2 years, whereas treatment with lenalidomide and dexamethasone will be continued.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed symptomatic MM based on either standard CRAB criteria (at least 10% of clonal bone marrow plasma cells plus CRAB defined as the onset of any of the following clinical symptoms: hypercalcemia, renal failure, anemia and bone lesions) or at least 10% of bone marrow plasma cells plus the presence of at least one of the following biomarkers of malignancy:

  * 60% or greater clonal plasma cells on bone marrow examination;
  * Serum involved/uninvolved free light chain (FLC) ratio of 100 or greater;
  * More than one focal lesion on magnetic resonance imaging (MRI) that is at least 5 mm or greater in size.
* Patient not eligible for ASCT (age ≥ 65 years or abnormal cardiac, pulmonary and liver function).
* Patient defined as fit or intermediate according to the IMWG (International Myeloma Working Group) frailty score
* Patient has given voluntary written informed consent.
* Patient is able to be compliant with hospital visits and procedures required per protocol.
* Patient agrees to use acceptable methods for contraception.
* Patient has measurable disease according to IMWG criteria.
* Patient has ECOG (Eastern Cooperative Oncology Group) performance status < 3.
* Pre-treatment clinical laboratory values within 30 days before randomization:

  * Platelet count ≥50 x 109/L (≥30 x 109 /L if myeloma involvement in the bone marrow is > 50%)
  * Absolute neutrophil count (ANC) ≥ 1 x 109/L without the use of growth factors
  * Corrected serum calcium ≤14 mg/dL (3.5 mmol/L)
  * Alanine transaminase (ALT): ≤ 3 x the ULN
  * Total bilirubin: ≤ 2 x the ULN
  * Calculated or measured creatinine clearance: ≥ 30 mL/minute.
* LVEF≥ 40%: 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation; multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available
* Pre-treatment blood pressure value < 140/90 mmHg even with adequate therapy: 24 hours blood pressure monitoring is the preferred method of evaluation; blood pressure diary at home for 2 weeks is acceptable.
* Females of childbearing potential (FBCP) comply with the conditions of the Pregnancy Prevention Plan, including confirmation that she has an adequate level of understanding.
* FBCP must follow the Pregnancy Prevention Plan and use a highly effective and an additional barrier contraception method simultaneously for 4 weeks before starting therapy, during treatment and dose interruptions and for at least 30 days after the last dose of study drugs*
* Males must use an effective barrier method of contraception if sexually active with FCBP during the treatment and for at least 90 days after the last administration of study drug/s. Male subjects must agree to refrain from sperm donation for at least 90 days after the last dose of carfilzomib.

Exclusion Criteria:

* Serious medical condition, laboratory abnormality or psychiatric illness that prevented the subject from the screening or place the subject at unacceptable risk.
* Patient defined as frail according to the IMWG frailty score.
* Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid < to the equivalent of dexamethasone 40 mg/day for 4 days).
* Pregnant or lactating females.
* Presence of:

  * Clinical active infectious hepatitis type A, B, C or HIV
  * Acute active infection requiring antibiotics or infiltrative pulmonary disease
  * Pulmonary hypertension and interstitial lung disease
  * Uncontrolled arrhythmias or history of QT prolongation
  * Myocardial infarction or unstable angina ≤ 6 months or other clinically significant heart disease
  * Peripheral neuropathy or neuropathic pain grade 2 or higher, as defined by National Cancer Institute Common Toxicity Criteria (NCI CTC) 5.0 (Appendix A)
  * Uncontrolled hypertension defined as persistent hypertension (>140/90 mmHg) regardless treatment with 3 drugs, including a diuretic.
* Contraindication to any of the required drugs or supportive treatments and hypersensitivity to any excipient of the study drugs.
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib).
* Invasive malignancy within the past 3 years.
* Administration of any experimental drug within 4 weeks prior the baseline or within 5 drug half-lives.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) | 5 years
  1. Minimal residual disease (MRD): unit of measure is not applicable, MRD is expressed as a pure number
Progression-free survival (PFS) | 5 years
  2. Progression-free survival (PFS): unit of measure is not applicable, PFS is expressed as a pure number

SECONDARY OUTCOMES:
Rate of drug reduction or drug discontinuation | 5 years
  Incidence of dose reduction and drug discontinuation in both treatment arms.
Cardiovascular assessment | 5 years
  Benefit of proper cardiovascular baseline assessment and monitoring during treatment in both treatment arms:to mitigate major cardiovascular adverse event incidence, to prolong duration of treatment, to improve efficacy.
Rate of dose reduction, drug discontinuation and toxicities | 5 years
  Safety as rate of dose reduction, drug discontinuation and toxicities
Response rate | 5 years
  Response rate will include complete response (CR), very good partial response (VGPR) and partial response (PR) using the International Response Criteria. Responders are defined as subjects with at least a PR.
Progression-free survival 2 (PFS2) | 5 years
  Time from randomization to objective tumor progression on next-line treatment or death from any cause.
Time to progression (TTP) | 5 years
  Time to progression will be measured from the date of randomization to the date of first observation of PD, or deaths related to PD.
Duration of response (DOR) | 5 years
  Time between first documentation of response and PD. Responders without disease progression will be censored either at the time of lost to FU, at the time of death due to other cause than PD, or at the end of the study.
Overall survival (OS) | 5 years
  Time between randomization and death. Subjects who die will be censored at time of death as an event, regardless cause of death.
Time to next therapy (TNT) | 5 years
  Time to next therapy will be measured from the date of randomization to the date of next anti-myeloma therapy. Death due to any cause before starting therapy will be considered an event.
MRD negativity | 5 years
  Correlation between MRD negativity and PFS, PFS2, TTP, TNT and OS
Prognostic factors | 5 years
  The following outcomes will be analysed in subgroups with different prognostic factors:
  * Progression-free survival (PFS),
  * Time to second disease progression (PFS2),
  * Time to progression (TTP),
  * Time to next therapy (TNT ),
  * Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bringhen, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (40):
- Italy (40):
  - AO "SS. Antonio e Biagio", Alessandria
  - AOU Ospedali Riuniti Umberto I, Ancona
  - Ospedale Mazzoni, Ascoli Piceno
  - Policlinico di Bari, Bari
  - Ospedali Riuniti, Bergamo
  - Azienda Sanitaria di Bolzano - Ospedale Lorenz B:Ohler, Bolzano
  - A.O. Spedali Civili di Brescia, Brescia
  - Ospedale "A. Businco", Cagliari
  - Istituto per la Cura e la RIcerca del Cancro di Candiolo, Candiolo
  - Ospedale Civico S. Croce e Carle, Cuneo
  - AOU Careggi, Florence
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola
  - Azienda Ospedaliera Papardo, Messina
  - Policlinico Universitario di Messina, Messina
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Europeo Oncologico, Milan
  - Istituto Nazionale Tumori, Milan
  - Ospedale Maggiore Policlinico di Milano, Milan
  - Università Federico II-Policlinico, Napoli
  - Ospedale Maggiore, Novara
  - AO San Luigi Gonzaga, Orbassano
  - AO di Padova, Padua
  - AO Cervello, Palermo
  - Ospedale S. Maria della Misericordia, Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - AO Bianchi Melacrino Morelli, Reggio Calabria
  - Ausl-Irccs, Reggio Emilia
  - Ospedale Infermi, Rimini
  - Ospedale Oncologico Regionale, Rionero in Vulture
  - ASL Roma 1, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - Ospedale S. Eugenio - Università Tor Vergata, Roma
  - Ospedale San Camillo Forlanini, Roma
  - Policlinico Umberto I - Università La Sapienza, Roma
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - AO S. Maria, Terni
  - AOU Città della Salute e della Scienza di Torino - PO Molinette - Ematologia U, Torino
  - AOU Città della Salute e della Scienza di Torino - PO Molinette, Torino
  - Policlinico Universitario di Udine, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bringhen S, Cani L, Antonioli E, Derudas D, Fazio F, Larocca A, Ronconi S, Cellini C, Falcone AP, Accardi F, Liberati AM, Galieni P, Belotti A, Cafro AM, Ria R, Benevolo G, Vincelli ID, Mannina D, Lotti F, Bruno B, Marasco V, Mazza R, Tosi P, Rivolti E, Boccadoro M, D'Agostino M. Carfilzomib-lenalidomide-dexamethasone versus lenalidomide-dexamethasone in patients with newly diagnosed myeloma ineligible for autologous stem-cell transplantation (EMN20): a randomised, open-label, multicentre, phase 3 trial. Lancet Haematol. 2025 Aug;12(8):e621-e634. doi: 10.1016/S2352-3026(25)00162-0. PMID 40769686